CLINICAL TRIAL: NCT05526443
Title: Austrian Registry for Evaluation of Treatment Patterns and Outcome in Patients With Advanced Pancreatic Ductal Adenocarcinoma (PDAC)
Acronym: ADPACA
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: ADPACA
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer; Advanced Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with locally advanced inoperable and/or metastatic pancreatic ductal adenocarcinoma: Patient with locally advanced inoperable and/or metastatic pancreatic ductal adenocarcinoma
  Interventions: Drug: all approved chemotherapeutic agents from second line

INTERVENTIONS:
Drug: all approved chemotherapeutic agents from second line — all approved chemotherapeutic agents from second line

SUMMARY:
To systematically collect and analyse real-world data on treatment patterns, clinical outcomes and toxicities among patients with advanced pancreatic ductal adenocarcinoma (PDAC) undergoing systematic treatment in Austria

DETAILED DESCRIPTION:
1500 adult patients with locally advanced inoperable and/or metastasized PDAC undergoing first line chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* 18 years, female and male
* ECOG (Eastern Cooperative Oncology Group) Scale 0-2
* Diagnosis of histologically confirmed locally advanced inoperable and/or metastatic PDAC
* Patients undergoing palliative 1st line therapy with a platinum- or gemcitabine- based chemotherapy in case of previous (neo)adjuvant therapy also patients who receive nal-Irinotecan/5-FU/Leukovorin as palliative first line are eglible
* Signed informed consent for prospective patients, for retrospective cases no informed consent is required

Exclusion Criteria:

* Patients with locally advanced operable PDAC who do not receive palliative chemotherapy
* Patients with locally advanced borderline resectable PDAC who do not receive palliative chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1500 adult patients with locally advanced inoperable and/or metastasized PDAC undergoing first line therapy with a platinum- or gemcitabin- based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with locally advanced inoperable and/or metastatic PDAC undergoing palliative second line therapy after progression on first line chemotherapy | 24 months

SECONDARY OUTCOMES:
To identify prognostic and predictive features for treatment efficacy | 24 months
To identify prognostic and predictive features for clinical outcome | 24 months
To identify prognostic and predictive features for Neuropathy | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events according to the Common Terminology Criteria of Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Febrile Neuropathy | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Thrombocytopenia | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Anemia | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Nausea/Vomiting | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Skin toxicity | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for rash | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for mucositis | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Fatigue | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for Allergic reactions | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To identify prognostic and predictive features for all other Adverse Events | 24 months
  Relative frequency of Grade 3 and Grade 4 Adverse Events (CTCAE) will be documented
To investigate the effect of dose density on treatment efficacy of first- and second line therapy | 24 months
To investigate the effect of dose modifications on treatment efficacy of first- and second line therapy | 24 months
To perform a comparative effectiveness analysis of different palliative second line chemotherapy regimens | 24 months
To evaluate treatment behaviours after progression on palliative second line therapy | 24 months
To analyse efficacy of palliative third line therapy | 24 months
To analyse patterns of BRCA testing in real-world practice | 24 months
To analyse the impact of BRCA testing in real-world practice on treatment decisions | 24 months
To analyse the impact of BRCA testing in real-world practice on outcome | 24 months
Prevalence of primary tumor resection in patients with metastatic or locally advanced inoperable pancreatic cancer | 24 months
Prevalence of metastasectomy in patients with metastatic or locally advanced inoperable pancreatic cancer | 24 months
To evaluate the impact of primary tumor resection on outcome | 24 months
To evaluate the impact of metastasectomy on outcome | 24 months
To evaluate the impact of primary granulocyte-colony stimulating factor (G-CSF) use on dose density of FOLFIRINOX | 24 months
To evaluate the impact of primary granulocyte-colony stimulating factor (G-CSF) use on rate of febrile neutropenia | 24 months
To evaluate the impact of primary granulocyte-colony stimulating factor (G-CSF) use on overall outcome | 24 months
To evaluate patterns of molecular profiling in the real world treatment practice of advanced pancreatic cancer | 24 months
To evaluate patterns of next generation sequencing (NGS) in the real world treatment practice of advanced pancreatic cancer | 24 months
To analyse treatment patterns and outcome in the subgroup of very young (<40 years old) patients with advanced pancreatic cancer | 24 months
To analyse treatment patterns and outcome in the subgroup of very old (>75 years old) patients with advanced pancreatic cancer | 24 months
To investigate the impact of diabetes mellitus on treatment efficacy of palliative chemotherapy and disease outcome | 24 months
To investigate the impact of antidiabetic therapy on treatment efficacy of palliative chemotherapy and disease outcome | 24 months
To analyze the mutational landscape of advanced pancreatic cancer and its impact on treatment decision making and clinical outcome | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Riedl, Priv.Doz. Dr., Principal Investigator — Medical University of Graz
Locations (12):
- Austria (12):
  - Medical University Graz Department of Oncology, Graz, Styria
  - Ordensklinikum Linz, Linz, Upper Austria
  - Landesklinikum Amstetten, Amstetten
  - Landesklinikum Feldkirch, Feldkirch
  - Krankenhaus der Barmherzigen Brüder, Graz
  - Universitätsklinikum Innsbruck,, Innsbruck
  - Landesklinikum Klagenfurt, Klagenfurt
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Barmherzige Schwestern Krankenhaus Wien, Vienna
  - Pancreatic Cancer Unit des Comprehensive Cancer Center (CCC-PCU), Vienna
  - St. Josef Krankenhaus Wien, Vienna
  - Krankenhaus St. Vinzenz Zams, Zams

IPD SHARING:
Plan to Share IPD: No